CLINICAL TRIAL: NCT06693232
Title: The Effect of Mobile Micro-learning on Critical Care Nurses' Self-confidence, Motivation, and Stress After Cardiopulmonary Resuscitation
Brief Title: Mobile Micro-learning on Nurses' Self-confidence, Motivation, and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: mobile micro-learning
Record Dates: First submitted 2024-11-10; First posted 2024-11-18 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2024-11

CONDITIONS: Cardiopulmonary Arrest; Nurse's Role
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: One group will receive mobile micro-learning.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Micro-mobile learning (Other): Critical care nurses will assess before intervention for the three outcomes
  Interventions: Procedure: Mobile micro-learning

INTERVENTIONS:
Procedure: Mobile micro-learning — Mobile micro-learning intervention contains a 10-minute video about cardiopulmonary resuscitation to continuously improve their self-confidence, motivation and reduce their stress

SUMMARY:
Before and after effect of using mobile micro-learning on their self-confidence, motivation, and stress toward cardiopulmonary resuscitation.

DETAILED DESCRIPTION:
This study aims to determine the effect of mobile micro-learning on critical care nurses' self-confidence, motivation, and stress after cardiopulmonary resuscitation.

The current study will use three scales. Self-Confidence Scale, Cardiopulmonary Motivation Scale, and Post-Code Stress Scale.

Mobile micro-learning is used easily to access video-based learning tips for effective practice for cardiopulmonary resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Critical care nurses who have worked in the intensive care unit for more than one year.

Exclusion Criteria:

* Critical care nurses who have less than one year of experience.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Self-Confidence Scale | before and after intervention immediately, after two week and after one month
  It contains 12 items on a 5-point Likert scale (1 = not confident; 2 = hardly confident; 3 = confident; 4 = very confident; and 5 = extremely confident), with scores ranging between 12 and 60, with higher scores indicating more confidence.
Cardiopulmonary motivation | before and after intervention immediately, after two week and after one month
  This instrument examined eight dimensions, including facilitators of resuscitation (6 items), feeling of achievement (7 items), high chances of success (8 items), low chances of success (6 items), recognition and appreciation (6 items), accountability (4 items), perceived importance (3 items), and beliefs (3 items). The scale of the questionnaire was a five-point Likert scale. More specifically, the first three items were rated on a scale ranging from always to never (i.e. 5 = always, 4 = most of the time,3 = sometimes,2 = rarely, and 1 = never). Moreover, the remaining items were rated on a scale ranging from completely agree to 'neither agree nor disagree (i.e. 5 = I completely agree score, 4 = I agree, 3 = I disagree, 2 = I completely disagree, and 1 = neither agree nor disagree).
Post-Code Stress Scale | before and after intervention immediately, after two week and after one month
  It consist of 20 items, the 5-level Likert scale, where: 1-the claim does not apply to me, 2-the claim hardly applies to me, 3-I cannot decide whether the claim applies to me or not, 4-the claim often applies to me and 5-the claim is typical of me

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of nursing, Damanhūr, Capital City of Beheira Governorate
  - Faculty of nursing Damanhour university, Damanhūr

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catani L, Gugliotta L, Campanini E, Mangianti S, Gibellini D, Baravelli S, Vianelli N, Lemoli RM, Tura S. Megakaryocyte progenitors derived from bone marrow or G-CSF-mobilized peripheral blood CD34 cells show a distinct phenotype and responsiveness to interleukin-3 (IL-3) and PEG-recombinant human megakaryocyte growth and development factor (PEG-rHuMGDF). Br J Haematol. 1998 Jan;100(1):207-18. doi: 10.1046/j.1365-2141.1998.00511.x. PMID 9450813
- [Background] Can S, Durgun H, Dalcali BK. Effect of online communication skills training on effective communication and self-efficacy and self-regulated learning skills of nursing students: A randomized controlled study. Nurse Educ Pract. 2022 Aug;63:103371. doi: 10.1016/j.nepr.2022.103371. Epub 2022 May 25. PMID 35839589